CLINICAL TRIAL: NCT07345533
Title: EXPLORATORY STUDY OF THE MYHEARTSENTINEL SYSTEM, A CARDIAMETRICS MEDICAL DEVICE - ANALYSIS OF CARDIAC ELECTROPHYSIOLOGICAL AND MECHANICAL SIGNALS DURING A DECOMPENSATION/RECOMPENSATION EPISODE IN PATIENTS WITH HEART FAILURE IN THE HOSPITAL AND UPON DISCHARGE HOME
Brief Title: EXPLORATORY STUDY OF THE MYHEARTSENTINEL SYSTEM, A CARDIAMETRICS MEDICAL DEVICE
Acronym: ASEMC-DR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-0232
Record Dates: First submitted 2025-12-12; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard of care plus MYHEARTSENTINEL SYSTEM device (Experimental)
  Interventions: Device: MYHEARTSENTINEL SYSTEM cutaneous DEVICE

INTERVENTIONS:
Device: MYHEARTSENTINEL SYSTEM cutaneous DEVICE — MYHEARTSENTINEL SYSTEM cutaneous DEVICE

SUMMARY:
Background:

Chronic heart failure represents a major public health challenge, affecting approximately 64 million people worldwide and generating high costs in terms of mortality, frequent hospitalizations, and medical expenses. In France, this disease is expected to cause nearly 70,000 deaths and 181,000 hospital admissions in 2022. Current management, based on periodic consultations, fails to effectively prevent acute exacerbations, highlighting the importance of technological solutions such as remote monitoring.

Objective:

This study aims to demonstrate the value of regular monitoring of electrophysiological and mechanical cardiac signals and parameters in patients with chronic heart failure. Its goal is to build a database of signals from an external measuring device to identify parameters that evolve in relation to biological and/or hemodynamic changes and/or the patient's clinical status. The results of this study will enable the further development of an automated monitoring solution for heart failure patients to enable early detection and management of decompensation.

Materials and Methods:

A total of 70 patients diagnosed with chronic heart failure will be included, including 30 patients hospitalized for heart failure decompensation and 40 patients hospitalized for hemodynamic assessment. Electrophysiological and cardiac mechanical data will be collected using a skin-based measuring device. These data will then be correlated with biological and/or hemodynamic changes and/or the patient's clinical status. They will contribute to the training of an algorithm to detect the risk of decompensation.

Hypothesis Tested:

The study will test the hypothesis that regular, automated remote monitoring of the data collected during the study can identify the risk of decompensation. Ultimately, this approach could improve the management of heart failure by maintaining a state of balance, while reducing the mental burden on patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 90 years
* Affiliated with the social security system.
* Patients who have been informed of the study and have signed informed consent.
* Patients with heart failure and one of the following two criteria:

  * Hospitalized for hemodynamic assessment
  * Hospitalized in a cardiology unit (ICU or telemetry unit) for congestive decompensation of known heart failure defined by [8] minimal dyspnea at rest or during exercise AND an elevation of BNP > 400 µg/ml or NT-proBNP > 1600 µg/ml

Exclusion Criteria:

* Patient hospitalized for decompensated heart failure due to an infectious cause requiring antibiotic treatment
* Patient requiring intravenous inotropes within the last 24 hours
* Patient with ventricular arrhythmias or permanent AF
* ACS with ST+ complex complicated by heart failure
* Valvulopathy awaiting interventional management
* Pericardial constriction
* Pregnant or breastfeeding women
* Women of childbearing potential without effective contraception
* Patients under guardianship, curatorship, legal protection, or legal protection.
* Patients already enrolled in an interventional clinical trial that may impact the electrophysiological and cardiac mechanical measurements of the medical device under study. • Inability to position the sensor on the thoracic area of interest
* Patients with open wounds, recent scars, or skin infections at the intended SCOUT device placement site
* Patients suffering from dermatitis, eczema, psoriasis, or other skin conditions at the placement site.
* Physical or psychological inability of the patient or caregiver to use the digital medical telemonitoring device and/or its collection accessories, as determined by the physician wishing to include the patient in the medical telemonitoring project;
* Patient refusal to transmit the data necessary to monitor the effective use of the DMN and to obtain individualized or national real-life usage results;
* Patient refusal to receive therapeutic support.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
ECG modification (yes/no) | baseline
  Identification of parameters/indicators that vary in relation to biological and/or hemodynamic changes and/or the patient's clinical condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France